CLINICAL TRIAL: NCT02025608
Title: Autonomic Function and Cardiovascular Risk in Restless Legs Syndrome: AUTOREST, a Case-control Study and a Randomized, Double-blind, Placebo-controlled, Parallel-group, 4-week, Multicenter Study of 0.25mg Pramipexole vs. Placebo in Patients With RLS
Brief Title: Autonomic Function and Cardiovascular Risk in Restless Legs Syndrome
Acronym: AUTOREST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mauro Manconi (Other)
Collaborators: Insel Gruppe AG, University Hospital Bern (Other); Cardiocentro Ticino (Other)
Responsible Party: Sponsor-Investigator, Mauro Manconi, Dr. med., Ospedale Regionale di Lugano
Organization: Ospedale Regionale di Lugano (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: NSI.13.01; 320030_144007 (Other Grant/Funding Number: Swiss National Science Foundation)
Record Dates: First submitted 2013-12-23; First posted 2014-01-01 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Restless Legs Syndrome
Keywords: Restless legs syndrome
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Pramipexole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pramipexole (Experimental): Pramipexole, 0.25 mg, daily for 4 weeks
  Interventions: Drug: Pramipexole
- Placebo (Placebo Comparator): Placebo, daily for 4 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pramipexole
  Arms: Pramipexole
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to explore whether patients with restless legs syndrome (RLS) differ from healthy subjects in daytime and night time autonomic function and cardiovascular risk markers and whether 4 week treatment with pramipexole affects autonomic function and cardiovascular risk markers in patients with RLS.

ELIGIBILITY:
Inclusion Criteria (all participants):

* Willingness to participate and written informed consent
* Aged 30 to 65 years at the time of screening
* Body mass index (BMI) ≤ 30
* Unremarkable neurological and physical examination
* Unremarkable standard blood parameter according to local reference values

Additional Inclusion Criteria for Restless Legs Syndrome (RLS) Patients:

* RLS according to current standard international criteria
* RLS symptoms ≥ 2 times per week for ≥ 1 year and during the past 12 months.
* Either current international RLS severity scale (IRLS) ≥ 15 or current IRLS ≥ 10 and RLS symptoms ≥ 4 times per week during the past 3 months.

Exclusion Criteria (all participants):

* Pregnancy, or breast feeding at time of screening.
* Recent anaesthesia (last 3 months).
* Sleep related breathing disorders during nocturnal polysomnography:
* Current history of psychiatric disorders according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV).
* Life time history of any diagnosis of, medication or intervention for cardiovascular diseases.
* Current chronic treatment that may affect autonomic function.
* Any significant neurological disease or diagnosed metabolic diseases that may affect cardiovascular function and/or increase cardiovascular risk.
* Any unstable medical condition.
* Smoking > 5 cigarettes per day during the last 2 years.
* Work involving night shifts (22:00 - 06:00 h) during the past 2 years.
* Travel with > 6 time zone differences during the past 6 months.
* Participation in any other study involving investigational or marketed products concomitantly or within 3 months prior to the screening visit.
* Current participation in other clinical trials.

Additional Exclusion Criteria for RLS Patients

* Exposure to dopaminergic drugs > 12 months during life time and/or > 1 week during the past 3 months and/or current or during the past month.
* Exposure to other RLS relevant medication (such as opioids, antiepileptics, clonidine except hypnotics such as benzodiazepines) > 24 months during life time and/or > 1 week during the past 3 months and/or current intake.
* Intake of hypnotics (such as benzodiazepines) during the past month.
* Other significant sleep disorder except symptoms potentially related to RLS such as insomnia and daytime sleepiness.
* Any contraindication or known hypersensitivity to dopaminergic drugs.

Additional Exclusion Criteria for Control Subjects

* Any pharmacological treatment that may affect sleep and/or sleep related movement disorders during the last 3 months.
* Any clinically significant sleep disorders according to the International Classification of Sleep Disorders (ICSD)12.
* Increased daytime sleepiness as indicated by an Epworth Sleepiness Scale (ESS) score > 11.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-12; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Change in heart rate activations during sleep from baseline to 4 weeks | Baseline, Week 4
  Number and amplitude of periodic leg movements during sleep (PLMS) and non-PLMS related heart rate activations during stable nocturnal sleep

SECONDARY OUTCOMES:
Change in baroreflex from baseline to 4 weeks | Baseline, Week 4
  Baroreflex sensitivity and baroreflex gain derived from tilt table tes
Change in blood serum markers from baseline to 4 weeks | Baseline, Week 4
  Highly-sensitive C reactive protein (hsCRP), lipoprotein-associated phospholipase A2 (lP-PLA2), and oxidised low density lipoprotein (oxLDL)

OTHER OUTCOMES:
Change in chemoreflexes from baseline to 4 weeks | Baseline, Week 4
  Peripheral and central chemoreflex sensitivity derived from carbon dioxide (CO2) rebreathing test

CONTACTS AND LOCATIONS:
Overall Officials: Mauro Manconi, PhD, MD, Principal Investigator — Neurocenter of Southern Switzerland; Claudio L.A. Bassetti, MD, Principal Investigator — Department of Neurology, Inselspital
Locations (2):
- Switzerland (2):
  - Neurocenter of Southern Switzerland, Lugano, Canton Ticino
  - Department of Neurology, Inselspital, Bern